CLINICAL TRIAL: NCT00274807
Title: Intensive Induction for Newly Diagnosed Acute Myelogenous Leukemia
Brief Title: Combination Chemotherapy in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Matt Kalaycio, Cleveland Clinic Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE-CCF-4409; P30CA043703 (NIH); CASE-CCF-4409; CASE-CCF-0645
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities | interventions — Filgrastim; Cytarabine; Etoposide; Mitoxantrone

INTERVENTIONS:
Biological: filgrastim
Drug: cytarabine
Drug: etoposide
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as mitoxantrone, cytarabine, and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying how well combination chemotherapy works in treating patients with newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete remission rate in patients with acute myelogenous leukemia treated with induction chemotherapy comprising mitoxantrone hydrochloride, cytarabine, and etoposide.
* Determine the feasibility and toxicity of this regimen when given to patients with newly diagnosed acute myelogenous leukemia.

OUTLINE: Patients receive induction chemotherapy comprising mitoxantrone hydrochloride IV on days 1-3, cytarabine IV continuously over 72 hours on days 1-3 and 8-10, and etoposide IV continuously over 72 hours on days 8-10. Patients also receive filgrastim (G-CSF) subcutaneously once daily beginning on day 4 and continuing until blood counts recover.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia

  * Previously untreated disease

    * Previous hydroxyurea and/or corticosteroids are acceptable
* No preexisting history of a hematologic disorder

  * Myelodysplastic features allowed
* No acute leukemia secondary to previous therapy
* No leukemic meningitis

PATIENT CHARACTERISTICS:

* Bilirubin < 2.0 mg/dL (unless felt to be increased because of hepatic infiltration with leukemia)
* Creatinine < 2.0 mg/dL
* Pregnant or lactating patients are ineligible
* Fertile patients must use effective contraception
* No history of or active congestive heart failure

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-06; Primary Completion 2007-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt E. Kalaycio, MD, Study Chair — The Cleveland Clinic